CLINICAL TRIAL: NCT07086313
Title: A Phase 2/3, Multicenter, Randomized, Double-blind, Placebo-controlled, Japan-China Joint Trial to Evaluate the Efficacy and Safety of Two Dose Levels of EB-1020 QD XR Capsules Administered Orally Once Daily in Children and Adolescents With Attention-deficit/Hyperactivity Disorder
Brief Title: A Trial to Evaluate the Efficacy and Safety of EB-1020 in Pediatric Patients With ADHD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 405-102-00114
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Attention-Deficit Hyperactivity Disorder(ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EB-1020(QD XR capsules) low dose (Experimental)
  Interventions: Drug: EB-1020 (Centanafadine) low dose
- EB-1020(QD XR capsules) high dose (Experimental)
  Interventions: Drug: EB-1020 (Centanafadine) high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EB-1020 (Centanafadine) low dose — low dose, capsule, oral, once daily, for 6 weeks
  Arms: EB-1020(QD XR capsules) low dose
Drug: EB-1020 (Centanafadine) high dose — high dose, capsule, oral, once daily, for 6 weeks
  Arms: EB-1020(QD XR capsules) high dose
Drug: Placebo — Placebo, capsule, oral, once daily, for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and examine the safety of two doses of EB-1020 QD XR capsule administered once daily orally in pediatric ADHD patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a primary diagnosis of ADHD based on DSM-5 diagnostic criteria, differentiated from other mental disorders using the MINI-KID, excluding other specified ADHD or unspecified ADHD.
* Participants with a symptom total raw score of>=28 (if not receiving any pharmacological treatment for ADHD) or>=22 (if receiving pharmacological treatment for ADHD) on the ADHD Rating Scale Version 5 (ADHD-RS-5) at screening.
* Participants with a symptom total raw score of>=28 on the ADHD-RS-5 at baseline.
* Participants with a score of 4 or higher on the Clinical Global Impression Severity - ADHD (CGI-S-ADHD) at baseline.

Exclusion Criteria:

* Participants who have a positive pregnancy test result at baseline.
* Participants determined to have the following diseases based on an interview using the MINI-KID.

  * Tourette's disorder
  * Panic disorder
  * Conduct disorder
  * Psychotic disorder
  * Post-traumatic stress disorder
  * Bipolar disorder
* Participants with a generalized anxiety disorder requiring pharmacotherapy, based on the DSM-5 diagnostic criteria.
* Participants with an autism spectrum disorder based on the DSM-5 diagnostic criteria.
* Participants with a personality disorder, oppositional defiant disorder, or obsessive-compulsive disorder that is the primary focus of treatment, based on the DSM-5 diagnostic criteria.
* Participants with a diagnosis of major depressive disorder (MDD), based on the DSM-5 diagnostic criteria who currently have a major depressive episode, or who have required treatment for MDD within the past 3 months prior to screening.

Also, participants who, in the judgment of the investigator or subinvestigator, may have a worsening of MDD during the trial or may require treatment during the trial period.

* Participants who have a diagnosis of intellectual disability with an intelligence quotient (IQ) score less than 70.
* Participants who have a significant risk of committing suicide in the opinion of the investigator or subinvestigator, or based on the following evidence.

  * Active suicidal ideation as evidenced by an answer of "yes" on Questions 4 or 5 (over the last 6 months) on the section of suicidal ideation or a history of suicidal behavior (over the last 6 months) on the Baseline/Screening version of the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening.
* Participants with a diagnosis of substance use disorder.

  * Platelets <= 130,000/mm3
  * Hemoglobin <= 11.2 g/dL
  * Neutrophils, absolute <= 1000/mm3
  * AST > 2 x ULN
  * ALT > 2 x ULN
  * eGFR < 45 mL/min/1.73 m2, calculated by the CKiD U25 equation
  * CPK >= 2 x ULN (except for the cases that the medical monitor determined that participant's inclusion is possible based on the discussion about the participant's condition with the investigator or subinvestigator)
  * Abnormal values for both free T4 and TSH
* Participants who cannot agree to discontinuation of prohibited concomitant medication, such as ADHD medication or antidepressants.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 315 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ADHD-RS-5 symptom total raw score at Week 6. | Baseline, Weeks 6
  The ADHD-RS-5 is an 18-item clinician rating scale to evaluate individual ADHD symptoms on a scale of 0 (never to rarely/no problem) to 3 (very often/severe problem). The total sum ranges from 0 (no ADHD symptoms) to 54 (extremely severe ADHD symptoms). Negative change from Baseline indicates improvement. Mixed-effect model repeated measure (MMRM) was used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Hokkaido University Hospital, Sapporo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.